CLINICAL TRIAL: NCT02531373
Title: A Phase I-II, Randomized, Double-Blind, Study to Evaluate the Safety, Tolerability, and Immunogenicity of Different Formulations of V114 in Healthy Adults and Infants
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of V114 in Healthy Adults and Infants (V114-005)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-005
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Adult: V114 Medium Dose (Experimental): Adult participants will receive a single 0.5 mL intramuscular injection of medium-dose V114 on Day 1.
  Interventions: Biological: V114 Medium Dose
- Adult: V114 High Dose (Experimental): Adult participants will receive a single 0.5 mL intramuscular injection of high-dose V114 on Day 1.
  Interventions: Biological: V114 High Dose
- Adult: V114 Medium Dose with Alternative Carrier Protein (Experimental): Adult participants will receive a single 0.5 mL intramuscular injection of medium-dose V114 with alternative carrier protein on Day 1.
  Interventions: Biological: V114 Medium Dose with Alternative Carrier Protein
- Adult: V114 High Dose with Alternative Carrier Protein (Experimental): Adult participants will receive a single 0.5 mL intramuscular injection of high-dose V114 with alternative carrier protein on Day 1.
  Interventions: Biological: V114 High Dose with Alternative Carrier Protein
- Infant: V114 Medium Dose (Experimental): Infant participants will receive a 0.5 mL intramuscular injection of medium-dose V114 at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 Medium Dose
- Infant: V114 High Dose (Experimental): Infant participants will receive a 0.5 mL intramuscular injection of high-dose V114 at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 High Dose
- Infant: V114 Medium Dose with Alternative Carrier Protein (Experimental): Infant participants will receive a 0.5 mL intramuscular injection of medium-dose V114 with alternative carrier protein at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 Medium Dose with Alternative Carrier Protein
- Infant: V114 High Dose with Alternative Carrier Protein (Experimental): Infant participants will receive a 0.5 mL intramuscular injection of high-dose V114 with alternative carrier protein at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 High Dose with Alternative Carrier Protein
- Infant: Prevnar 13™ (Active Comparator): Infant participants will receive a 0.5 mL intramuscular injection of Prevnar 13™ at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: Prevnar 13™

INTERVENTIONS:
Biological: V114 Medium Dose — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and Merck Aluminum Phosphate Adjuvant (125 mcg) in each 0.5 mL dose
  Arms: Adult: V114 Medium Dose; Infant: V114 Medium Dose
Biological: V114 High Dose — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (4 mcg each), serotype 6B (8 mcg), and Merck Aluminum Phosphate Adjuvant (250 mcg) in each 0.5 mL dose
  Arms: Adult: V114 High Dose; Infant: V114 High Dose
Biological: V114 Medium Dose with Alternative Carrier Protein — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg), and Merck Aluminum Phosphate Adjuvant (125 mcg) with alternative carrier protein in each 0.5 mL dose
  Arms: Adult: V114 Medium Dose with Alternative Carrier Protein; Infant: V114 Medium Dose with Alternative Carrier Protein
Biological: V114 High Dose with Alternative Carrier Protein — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (4 mcg each), serotype 6B (8 mcg), and Merck Aluminum Phosphate Adjuvant (250 mcg) with alternative carrier protein in each 0.5 mL dose
  Arms: Adult: V114 High Dose with Alternative Carrier Protein; Infant: V114 High Dose with Alternative Carrier Protein
Biological: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg) in each 0.5 ml dose
  Arms: Infant: Prevnar 13™

SUMMARY:
This study is designed to assess the effect of different dose levels of pneumococcal polysaccharide and adjuvant on the safety and immunogenicity of V114 in healthy adults and infants.

ELIGIBILITY:
Inclusion Criteria:

Adult Cohort: 18 to 49 years and in good health

* Highly unlikely to conceive from vaccination through 6 weeks after administration of the study vaccine.

Infant Cohort: approximately 2 months (42 to 90 days) and in good health.

Exclusion Criteria:

Adult cohort: Prior administration of any pneumococcal vaccine

* History of invasive pneumococcal disease
* Known hypersensitivity to any vaccine component
* Known or suspected impairment of immune function
* Coagulation disorder contraindicating intramuscular vaccination
* Received a blood transfusion or blood products within 6 months
* Participated in another clinical study of an investigational product within 2 months
* Breast feeding. Infant cohort: Prior administration of any pneumococcal vaccine
* Known hypersensitivity to any vaccine component
* Known or suspected impairment of immune function
* History of congenital or acquired immunodeficiency
* Has or mother has documented Human Immunodeficiency virus (HIV) infection
* Has or mother has documented hepatitis B surface antigen positive result
* Functional or anatomic asplenia
* History of failure to thrive
* Coagulation disorder contraindicating intramuscular vaccination
* History of autoimmune disease or autoimmune disorder
* Known neurologic or cognitive behavioral disorder
* Received systemic corticosteroids within 14 days
* Received other licensed non-live vaccine within 14 days
* Received other licensed live virus vaccine within 30 days
* Received a blood transfusion or blood products
* Participated in another clinical study of an investigational product
* History of invasive pneumococcal disease

Ages: 2 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 338 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rupp R, Hurley D, Grayson S, Li J, Nolan K, McFetridge RD, Hartzel J, Abeygunawardana C, Winters M, Pujar H, Benner P, Musey L. A dose ranging study of 2 different formulations of 15-valent pneumococcal conjugate vaccine (PCV15) in healthy infants. Hum Vaccin Immunother. 2019;15(3):549-559. doi: 10.1080/21645515.2019.1568159. Epub 2019 Feb 15. PMID 30689507

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults: V114 Medium Dose: Adult participants received a single 0.5 mL intramuscular injection of medium-dose V114 on Day 1
- Adults: V114 High Dose: Adult participants received a single 0.5 mL intramuscular injection of high-dose V114 on Day 1
- Adults: V114 Medium Dose + ACP: Adult participants received a single 0.5 mL intramuscular injection of medium-dose V114 with alternative carrier protein (ACP) on Day 1
- Adults: V114 High Dose + ACP: Adult participants received a single 0.5 mL intramuscular injection of high-dose V114 with ACP on Day 1
- Infants: V114 Medium Dose: Infant participants received a single 0.5 mL intramuscular injection of medium-dose V114 at 2, 4, 6, and 12-15 months of age
- Infants: V114 High Dose: Infant participants received a single 0.5 mL intramuscular injection of high-dose V114 at 2, 4, 6, and 12-15 months of age
- Infants: V114 Medium Dose + ACP: Infant participants received a single 0.5 mL intramuscular injection of medium-dose V114 with alternative carrier protein (ACP) at 2, 4, 6, and 12-15 months of age
- Infants: V114 High Dose + ACP: Infant participants received a single 0.5 mL intramuscular injection of high-dose V114 with ACP at 2, 4, 6, and 12-15 months of age
- Infants: Prevnar 13™: Infant participants received a single 0.5 mL intramuscular injection of Prevnar 13™ at 2, 4, 6, and 12-15 months of age
Period: Overall Study
Arm/Group | Adults: V114 Medium Dose | Adults: V114 High Dose | Adults: V114 Medium Dose + ACP | Adults: V114 High Dose + ACP | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: V114 Medium Dose + ACP | Infants: V114 High Dose + ACP | Infants: Prevnar 13™
Started | 20 | 20 | 20 | 20 | 51 | 51 | 52 | 52 | 52
Vaccination 1 | 20 | 20 | 20 | 20 | 50 | 50 | 52 | 52 | 52
Vaccination 2 | 0 | 0 | 0 | 0 | 49 | 48 | 50 | 51 | 51
Vaccination 3 | 0 | 0 | 0 | 0 | 48 | 47 | 49 | 51 | 49
Vaccination 4 | 0 | 0 | 0 | 0 | 44 | 43 | 43 | 43 | 43
Completed | 20 | 20 | 20 | 20 | 43 | 42 | 41 | 43 | 43
Not Completed | 0 | 0 | 0 | 0 | 8 | 9 | 11 | 9 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 8 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one study vaccination
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults: V114 Medium Dose | Adults: V114 High Dose | Adults: V114 Medium Dose + ACP | Adults: V114 High Dose + ACP | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: V114 Medium Dose + ACP | Infants: V114 High Dose + ACP | Infants: Prevnar 13™ | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 50 | 50 | 52 | 52 | 52 | 336
Age, Customized [Count of Participants; unit: Participants]
  6 weeks | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 3 | 1 | 9
  7 weeks | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 4 | 2 | 15
  8 weeks | 0 | 0 | 0 | 0 | 19 | 15 | 16 | 19 | 26 | 95
  9 weeks | 0 | 0 | 0 | 0 | 14 | 22 | 22 | 20 | 16 | 94
  10 weeks | 0 | 0 | 0 | 0 | 4 | 6 | 4 | 4 | 2 | 20
  11 weeks | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 0 | 4 | 16
  12 weeks | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 7
  18 to 29 years | 6 | 4 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 20
  30 to 39 years | 10 | 9 | 10 | 6 | 0 | 0 | 0 | 0 | 0 | 35
  40 to 49 years | 4 | 7 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 11 | 13 | 23 | 23 | 29 | 32 | 25 | 182
  Male | 8 | 6 | 9 | 7 | 27 | 27 | 23 | 20 | 27 | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 3 | 4 | 2 | 3 | 7 | 6 | 5 | 8 | 7 | 45
  White | 14 | 16 | 18 | 16 | 38 | 40 | 41 | 41 | 40 | 264
  More than one race | 3 | 0 | 0 | 0 | 5 | 3 | 5 | 3 | 5 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adults: Percentage of Participants With an Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 6 weeks after vaccination
Population: The analysis population included all randomized adult participants who received study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults: V114 Medium Dose | Adults: V114 High Dose | Adults: V114 Medium Dose + ACP | Adults: V114 High Dose + ACP
Number analyzed (Participants) | 20 | 20 | 20 | 20
Percentage of participants | 90.0 [68.3 to 98.8] | 95.0 [75.1 to 99.9] | 95.0 [75.1 to 99.9] | 95.0 [75.1 to 99.9]

2. Primary Outcome: Infants: Percentage of Participants With an Adverse Event
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 1 month after Vaccination 4 (Month 11-15)
Population: The analysis population included all randomized infant participants who received at least one dose of study vaccination. One cross-treated participant in the Infants: V114 Medium Dose + ACP group was excluded from the safety analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: V114 Medium Dose + ACP | Infants: V114 High Dose + ACP | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 51 | 52 | 52
Percentage of participants | 96.0 | 94.0 | 96.1 | 98.1 | 100.0
Statistical Analysis 1: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = -4.0, 95% CI 2-sided [-13.5 to 3.1]
Statistical Analysis 2: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = -6.0, 95% CI 2-sided [-16.3 to 1.2]
Statistical Analysis 3: Comparison: Infants: V114 Medium Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = -3.9, 95% CI 2-sided [-13.3 to 3.2]
Statistical Analysis 4: Comparison: Infants: V114 High Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = -1.9, 95% CI 2-sided [-10.2 to 5.1]

3. Primary Outcome: Infants: Percentage of Participants With Study Vaccination Withdrawn Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to time of Vaccination 4 (Month 10-13)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: V114 Medium Dose + ACP | Infants: V114 High Dose + ACP | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 51 | 52 | 52
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-6.9 to 7.2]
Statistical Analysis 2: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-6.9 to 7.2]
Statistical Analysis 3: Comparison: Infants: V114 Medium Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-6.9 to 7.1]
Statistical Analysis 4: Comparison: Infants: V114 High Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-6.9 to 6.9]

4. Primary Outcome: Infants: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: Solicited injection-site AEs were injection-site erythema, injection-site induration, injection-site pain, and injection-site swelling.
Time Frame: Up to 14 days after any vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: V114 Medium Dose + ACP | Infants: V114 High Dose + ACP | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 51 | 52 | 52
Percentage of participants | 78.0 | 80.0 | 58.8 | 80.8 | 57.7
Statistical Analysis 1: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.029, Miettinen and Nurminen method; Risk Difference (RD) = 20.3, 95% CI 2-sided [2.1 to 37.3]
Statistical Analysis 2: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.016, Miettinen and Nurminen method; Risk Difference (RD) = 22.3, 95% CI 2-sided [4.3 to 39.1]
Statistical Analysis 3: Comparison: Infants: V114 Medium Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.908, Miettinen and Nurminen method; Risk Difference (RD) = 1.1, 95% CI 2-sided [-17.7 to 19.9]
Statistical Analysis 4: Comparison: Infants: V114 High Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.011, Miettinen and Nurminen method; Risk Difference (RD) = 23.1, 95% CI 2-sided [5.4 to 39.6]

5. Primary Outcome: Infants: Percentage of Participants With a Solicited Systemic Adverse Event
Description: Solicited systemic AEs were irritability, decreased appetite, somnolence, and urticaria.
Time Frame: Up to 14 days after any vaccination
Population: The analysis population included all randomized infant participants who received at least one dose of study vaccination and had follow-up for the outcome measure. One cross-treated participant in the Infants: V114 Medium Dose + ACP group was excluded from the safety analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: V114 Medium Dose + ACP | Infants: V114 High Dose + ACP | Infants: Prevnar 13™
Number analyzed (Participants) | 44 | 43 | 47 | 49 | 46
Percentage of participants | 88.0 | 86.0 | 92.2 | 94.2 | 88.5
Statistical Analysis 1: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.943, Miettinen and Nurminen method; Risk Difference (RD) = -0.5, 95% CI 2-sided [-14.0 to 12.9]
Statistical Analysis 2: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.711, Miettinen and Nurminen method; Risk Difference (RD) = -2.5, 95% CI 2-sided [-16.4 to 11.2]
Statistical Analysis 3: Comparison: Infants: V114 Medium Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.529, Miettinen and Nurminen method; Risk Difference (RD) = 3.7, 95% CI 2-sided [-8.7 to 16.4]
Statistical Analysis 4: Comparison: Infants: V114 High Dose + ACP vs Infants: Prevnar 13™; Test type: Equivalence — Miettinen and Nurminen method; p = 0.298, Miettinen and Nurminen method; Risk Difference (RD) = 5.8, 95% CI 2-sided [-5.8 to 18.2]

6. Primary Outcome: Infants: Geometric Mean Concentration (GMC) of Pneumococcal Serotype IgG Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: 1 month after Vaccination 3 (Month 5)
Population: The analysis population included all infant participants who did not have a protocol violation that could have impacted the validity of the antibody responses. This outcome measure was exploratory for the groups receiving ACP-containing vaccine; results for those groups are thus not included here.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 52
µg/mL
  Serotype 1: number analyzed (Participants) | 37 | 39 | 40
  Serotype 1 | 1.33 [1.07 to 1.67] | 1.49 [1.19 to 1.87] | 1.63 [1.28 to 2.07]
  Serotype 3: number analyzed (Participants) | 37 | 39 | 40
  Serotype 3 | 0.94 [0.78 to 1.13] | 1.12 [0.89 to 1.41] | 0.53 [0.42 to 0.67]
  Serotype 4: number analyzed (Participants) | 37 | 39 | 40
  Serotype 4 | 1.46 [1.20 to 1.77] | 1.31 [1.05 to 1.64] | 1.14 [0.89 to 1.45]
  Serotype 5: number analyzed (Participants) | 37 | 39 | 40
  Serotype 5 | 1.29 [0.96 to 1.74] | 1.13 [0.83 to 1.55] | 1.36 [0.94 to 1.98]
  Serotype 6A: number analyzed (Participants) | 37 | 39 | 40
  Serotype 6A | 1.41 [0.95 to 2.10] | 1.52 [1.07 to 2.16] | 2.82 [1.93 to 4.12]
  Serotype 6B: number analyzed (Participants) | 37 | 39 | 40
  Serotype 6B | 1.80 [1.15 to 2.82] | 1.30 [0.83 to 2.02] | 1.62 [1.01 to 2.61]
  Serotype 7F: number analyzed (Participants) | 37 | 39 | 40
  Serotype 7F | 2.23 [1.77 to 2.81] | 2.87 [2.44 to 3.37] | 2.97 [2.24 to 3.93]
  Serotype 9V: number analyzed (Participants) | 37 | 39 | 40
  Serotype 9V | 1.68 [1.24 to 2.29] | 1.44 [1.05 to 1.97] | 1.48 [1.10 to 1.97]
  Serotype 14: number analyzed (Participants) | 37 | 39 | 40
  Serotype 14 | 4.24 [3.31 to 5.42] | 4.58 [3.70 to 5.67] | 4.94 [3.51 to 6.95]
  Serotype 18C: number analyzed (Participants) | 37 | 39 | 40
  Serotype 18C | 0.96 [0.71 to 1.31] | 1.22 [0.99 to 1.51] | 1.54 [1.14 to 2.07]
  Serotype 19A: number analyzed (Participants) | 37 | 39 | 40
  Serotype 19A | 1.47 [1.18 to 1.82] | 1.43 [1.19 to 1.72] | 1.63 [1.20 to 2.21]
  Serotype 19F: number analyzed (Participants) | 37 | 39 | 40
  Serotype 19F | 1.81 [1.44 to 2.28] | 2.37 [1.99 to 2.83] | 2.19 [1.80 to 2.66]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 37 | 39 | 40
  Serotype 22F (non-Prevnar serotype) | 4.34 [3.40 to 5.55] | 4.79 [3.88 to 5.91] | 0.05 [0.05 to 0.06]
  Serotype 23F: number analyzed (Participants) | 37 | 38 | 40
  Serotype 23F | 1.08 [0.72 to 1.62] | 1.16 [0.83 to 1.61] | 1.19 [0.82 to 1.71]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 37 | 39 | 40
  Serotype 33F (non-Prevnar serotype) | 1.32 [0.79 to 2.21] | 1.09 [0.64 to 1.85] | 0.06 [0.05 to 0.07]
Statistical Analysis 1: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 1; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.61 to 1.10]
Statistical Analysis 2: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 3; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 1.77, 95% CI 2-sided [1.33 to 2.35]
Statistical Analysis 3: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 4; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.91 to 1.81]
Statistical Analysis 4: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 5; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.59 to 1.51]
Statistical Analysis 5: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 6A; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.50, 95% CI [0.29 to 0.86]
Statistical Analysis 6: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 6B; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.58 to 2.10]
Statistical Analysis 7: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 7F; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.55 to 1.03]
Statistical Analysis 8: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 9V; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.74 to 1.75]
Statistical Analysis 9: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 14; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.58 to 1.27]
Statistical Analysis 10: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 18C; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.63, 95% CI [0.43 to 0.92]
Statistical Analysis 11: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 19A; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.64 to 1.26]
Statistical Analysis 12: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 19F; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.62 to 1.11]
Statistical Analysis 13: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 22F (non-Prevnar serotype); Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 81.47, 95% CI 2-sided [60.51 to 109.68]
Statistical Analysis 14: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 23F; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.56 to 1.47]
Statistical Analysis 15: Comparison: Infants: V114 Medium Dose vs Infants: Prevnar 13™; Serotype 33F (non-Prevnar serotype); Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 22.23, 95% CI 2-sided [11.77 to 41.97]
Statistical Analysis 16: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 1; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.68 to 1.23]
Statistical Analysis 17: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 3; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 2.11, 95% CI 2-sided [1.60 to 2.80]
Statistical Analysis 18: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 4; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.82 to 1.62]
Statistical Analysis 19: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 5; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.53 to 1.31]
Statistical Analysis 20: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 6A; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.54, 95% CI 2-sided [0.31 to 0.92]
Statistical Analysis 21: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 6B; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.42 to 1.50]
Statistical Analysis 22: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 7F; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.71 to 1.31]
Statistical Analysis 23: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 9V; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.64 to 1.49]
Statistical Analysis 24: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 14; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.63 to 1.37]
Statistical Analysis 25: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 18C; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.55 to 1.16]
Statistical Analysis 26: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 19A; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.63 to 1.22]
Statistical Analysis 27: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 19F; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.81 to 1.44]
Statistical Analysis 28: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 22F (non-Prevnar serotype); Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 89.87, 95% CI 2-sided [67.02 to 120.51]
Statistical Analysis 29: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 23F; Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.61 to 1.57]
Statistical Analysis 30: Comparison: Infants: V114 High Dose vs Infants: Prevnar 13™; Serotype 33F (non-Prevnar serotype); Test type: Equivalence — 2-sample t-test; Risk Ratio (RR) = 18.38, 95% CI 2-sided [9.82 to 34.41]

7. Secondary Outcome: Adults: Geometric Mean Concentration (GMC) of Pneumococcal Serotype IgG Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: 1 month after vaccination
Population: The analysis population included all adult participants who did not have a protocol violation that could have impacted the validity of the antibody responses. This outcome measure was exploratory for the groups receiving ACP-containing vaccine; results for those groups are thus not included here.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Adults: V114 Medium Dose | Adults: V114 High Dose
Number analyzed (Participants) | 20 | 20
µg/mL
  Serotype 1: number analyzed (Participants) | 20 | 18
  Serotype 1 | 3.47 [1.83 to 6.61] | 4.99 [2.51 to 9.93]
  Serotype 3: number analyzed (Participants) | 20 | 18
  Serotype 3 | 0.50 [0.31 to 0.82] | 0.71 [0.44 to 1.15]
  Serotype 4: number analyzed (Participants) | 20 | 18
  Serotype 4 | 0.96 [0.56 to 1.65] | 1.47 [0.76 to 2.86]
  Serotype 5: number analyzed (Participants) | 20 | 18
  Serotype 5 | 3.08 [1.41 to 6.74] | 2.20 [1.02 to 4.77]
  Serotype 6A: number analyzed (Participants) | 20 | 18
  Serotype 6A | 8.42 [3.55 to 19.98] | 4.78 [1.99 to 11.47]
  Serotype 6B: number analyzed (Participants) | 20 | 18
  Serotype 6B | 7.25 [3.03 to 17.35] | 3.71 [1.36 to 10.14]
  Serotype 7F: number analyzed (Participants) | 20 | 18
  Serotype 7F | 5.12 [2.35 to 11.17] | 6.12 [3.30 to 11.34]
  Serotype 9V: number analyzed (Participants) | 20 | 18
  Serotype 9V | 2.76 [1.18 to 6.46] | 2.27 [1.28 to 4.04]
  Serotype 14: number analyzed (Participants) | 20 | 18
  Serotype 14 | 14.97 [6.62 to 33.84] | 9.96 [4.24 to 23.41]
  Serotype 18C: number analyzed (Participants) | 20 | 18
  Serotype 18C | 9.48 [4.51 to 19.91] | 8.91 [4.40 to 18.04]
  Serotype 19A: number analyzed (Participants) | 20 | 18
  Serotype 19A | 15.19 [9.85 to 23.41] | 4.62 [2.61 to 8.16]
  Serotype 19F: number analyzed (Participants) | 20 | 18
  Serotype 19F | 8.67 [4.15 to 18.15] | 7.96 [4.33 to 14.61]
  Serotype 22F: number analyzed (Participants) | 20 | 18
  Serotype 22F | 2.93 [1.80 to 4.78] | 4.04 [2.38 to 6.86]
  Serotype 23F: number analyzed (Participants) | 20 | 18
  Serotype 23F | 11.55 [5.78 to 23.08] | 8.91 [4.14 to 19.20]
  Serotype 33F: number analyzed (Participants) | 20 | 18
  Serotype 33F | 4.06 [1.66 to 9.93] | 6.16 [3.18 to 11.94]

8. Secondary Outcome: Adults: Geometric Mean Fold Rise (GMFR) From Baseline in GMC of Pneumococcal Serotype IgG Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay. GMFR is defined as the geometric mean of the ratio of concentration at 1 month after vaccination divided by concentration at baseline.
Time Frame: Baseline and 1 month after vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Adults: V114 Medium Dose | Adults: V114 High Dose
Number analyzed (Participants) | 20 | 20
Ratio
  Serotype 1: number analyzed (Participants) | 20 | 18
  Serotype 1 | 14.94 [7.73 to 28.90] | 14.41 [7.93 to 26.17]
  Serotype 3: number analyzed (Participants) | 20 | 18
  Serotype 3 | 3.12 [2.08 to 4.67] | 4.73 [2.82 to 7.92]
  Serotype 4: number analyzed (Participants) | 20 | 18
  Serotype 4 | 7.24 [4.21 to 12.45] | 12.66 [6.20 to 25.86]
  Serotype 5: number analyzed (Participants) | 20 | 18
  Serotype 5 | 6.59 [3.31 to 13.12] | 5.79 [2.91 to 11.52]
  Serotype 6A: number analyzed (Participants) | 20 | 18
  Serotype 6A | 47.27 [23.68 to 94.36] | 23.26 [11.98 to 45.14]
  Serotype 6B: number analyzed (Participants) | 20 | 18
  Serotype 6B | 35.70 [17.46 to 73.00] | 18.23 [8.84 to 37.62]
  Serotype 7F: number analyzed (Participants) | 20 | 18
  Serotype 7F | 12.84 [6.71 to 24.56] | 17.51 [9.58 to 32.02]
  Serotype 9V: number analyzed (Participants) | 20 | 18
  Serotype 9V | 12.28 [5.37 to 28.10] | 14.61 [7.81 to 27.35]
  Serotype 14: number analyzed (Participants) | 20 | 18
  Serotype 14 | 14.99 [5.96 to 37.67] | 11.96 [5.80 to 24.64]
  Serotype 18C: number analyzed (Participants) | 20 | 18
  Serotype 18C | 29.41 [15.09 to 57.32] | 38.44 [18.66 to 79.20]
  Serotype 19A: number analyzed (Participants) | 20 | 18
  Serotype 19A | 8.04 [4.26 to 15.18] | 8.80 [5.12 to 15.14]
  Serotype 19F: number analyzed (Participants) | 20 | 18
  Serotype 19F | 20.63 [9.35 to 45.55] | 13.52 [6.49 to 28.19]
  Serotype 22F: number analyzed (Participants) | 20 | 18
  Serotype 22F | 12.87 [6.86 to 24.16] | 20.85 [11.81 to 36.82]
  Serotype 23F: number analyzed (Participants) | 20 | 18
  Serotype 23F | 45.59 [25.61 to 81.18] | 28.44 [16.04 to 50.44]
  Serotype 33F: number analyzed (Participants) | 20 | 18
  Serotype 33F | 9.69 [4.25 to 22.10] | 13.25 [6.07 to 28.92]

9. Secondary Outcome: Infants: Percentage of Participants With GMC ≥0.35 µg/mL at 1 Month After Vaccination 3
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: 1 month after Vaccination 3 (Month 5)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 52
Percentage of participants
  Serotype 1: number analyzed (Participants) | 37 | 39 | 40
  Serotype 1 | 97.3 [85.84 to 99.93] | 100.0 [90.97 to 100.0] | 100.0 [91.19 to 100.0]
  Serotype 3: number analyzed (Participants) | 37 | 39 | 40
  Serotype 3 | 94.6 [81.81 to 99.34] | 97.4 [86.52 to 99.94] | 70.0 [53.47 to 83.44]
  Serotype 4: number analyzed (Participants) | 37 | 39 | 40
  Serotype 4 | 100.0 [90.51 to 100.0] | 97.4 [86.52 to 99.94] | 95.0 [83.08 to 99.39]
  Serotype 5: number analyzed (Participants) | 37 | 39 | 40
  Serotype 5 | 94.6 [81.81 to 99.34] | 84.6 [69.47 to 94.14] | 85.0 [70.16 to 94.29]
  Serotype 6A: number analyzed (Participants) | 37 | 39 | 40
  Serotype 6A | 91.9 [78.09 to 98.30] | 89.7 [75.78 to 97.13] | 95.0 [83.08 to 99.39]
  Serotype 6B: number analyzed (Participants) | 37 | 30 | 40
  Serotype 6B | 89.2 [74.58 to 96.97] | 82.1 [66.47 to 92.46] | 85.0 [70.16 to 94.29]
  Serotype 7F: number analyzed (Participants) | 37 | 39 | 40
  Serotype 7F | 100.0 [90.51 to 100.0] | 100.0 [90.97 to 100.0] | 100.0 [91.19 to 100.0]
  Serotype 9V: number analyzed (Participants) | 37 | 39 | 40
  Serotype 9V | 94.6 [81.81 to 99.34] | 92.3 [79.13 to 98.38] | 95.0 [83.08 to 99.39]
  Serotype 14: number analyzed (Participants) | 37 | 30 | 40
  Serotype 14 | 100.0 [90.51 to 100.0] | 100.0 [90.97 to 100.0] | 97.5 [86.84 to 99.94]
  Serotype 18C: number analyzed (Participants) | 37 | 39 | 40
  Serotype 18C | 86.5 [71.23 to 95.46] | 97.4 [86.52 to 99.94] | 97.5 [86.84 to 99.94]
  Serotype 19A: number analyzed (Participants) | 37 | 39 | 40
  Serotype 19A | 94.6 [81.81 to 99.34] | 100.0 [90.97 to 100.0] | 95.0 [83.08 to 99.39]
  Serotype 19F: number analyzed (Participants) | 37 | 39 | 40
  Serotype 19F | 97.3 [85.84 to 99.93] | 100.0 [90.97 to 100.0] | 100.0 [91.19 to 100.0]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 37 | 39 | 40
  Serotype 22F (non-Prevnar serotype) | 100.0 [90.51 to 100.0] | 100.0 [90.97 to 100.0] | 0.0 [0.00 to 8.81]
  Serotype 23F: number analyzed (Participants) | 37 | 38 | 40
  Serotype 23F | 86.5 [71.23 to 95.46] | 86.8 [71.91 to 95.59] | 85.0 [70.16 to 94.29]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 37 | 39 | 40
  Serotype 33F (non-Prevnar serotype) | 81.1 [64.84 to 92.04] | 71.8 [55.13 to 85.00] | 0.0 [0.00 to 8.81]

10. Secondary Outcome: Infants: Percentage of Participants With GMC ≥0.35 µg/mL Before Vaccination 4
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: Before Vaccination 4 (Month 10-13)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 52
Percentage of participants
  Serotype 1: number analyzed (Participants) | 39 | 39 | 40
  Serotype 1 | 30.8 [17.02 to 47.57] | 43.6 [27.81 to 60.38] | 57.5 [40.89 to 72.96]
  Serotype 3: number analyzed (Participants) | 39 | 39 | 40
  Serotype 3 | 10.3 [2.87 to 24.22] | 15.4 [5.86 to 30.53] | 7.5 [1.57 to 20.39]
  Serotype 4: number analyzed (Participants) | 39 | 39 | 40
  Serotype 4 | 17.9 [7.54 to 33.53] | 33.3 [19.09 to 50.22] | 27.5 [14.60 to 43.89]
  Serotype 5: number analyzed (Participants) | 39 | 39 | 40
  Serotype 5 | 61.5 [44.62 to 76.64] | 56.4 [39.62 to 72.19] | 72.5 [56.11 to 85.40]
  Serotype 6A: number analyzed (Participants) | 39 | 39 | 40
  Serotype 6A | 48.7 [32.42 to 65.22] | 56.4 [39.62 to 72.19] | 82.5 [67.22 to 92.66]
  Serotype 6B: number analyzed (Participants) | 39 | 39 | 40
  Serotype 6B | 71.8 [55.13 to 85.00] | 71.8 [55.13 to 85.00] | 62.5 [45.80 to 77.27]
  Serotype 7F: number analyzed (Participants) | 39 | 39 | 40
  Serotype 7F | 82.1 [66.47 to 92.46] | 92.3 [79.13 to 98.38] | 97.5 [86.84 to 99.94]
  Serotype 9V: number analyzed (Participants) | 39 | 39 | 40
  Serotype 9V | 53.8 [37.18 to 69.91] | 64.1 [47.18 to 78.80] | 45.0 [29.26 to 61.51]
  Serotype 14: number analyzed (Participants) | 39 | 39 | 40
  Serotype 14 | 87.2 [72.57 to 95.70] | 87.2 [72.57 to 95.70] | 87.5 [73.20 to 95.81]
  Serotype 18C: number analyzed (Participants) | 39 | 39 | 40
  Serotype 18C | 12.8 [4.30 to 27.43] | 23.1 [11.13 to 39.33] | 35.0 [20.63 to 51.68]
  Serotype 19A: number analyzed (Participants) | 39 | 39 | 40
  Serotype 19A | 33.3 [19.09 to 50.22] | 28.2 [15.00 to 44.87] | 55.0 [38.49 to 70.74]
  Serotype 19F: number analyzed (Participants) | 39 | 39 | 40
  Serotype 19F | 35.9 [21.20 to 52.82] | 46.2 [30.09 to 62.82] | 62.5 [45.80 to 77.27]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 39 | 39 | 40
  Serotype 22F (non-Prevnar serotype) | 97.4 [86.52 to 99.94] | 97.4 [86.52 to 99.94] | 2.5 [0.06 to 13.16]
  Serotype 23F: number analyzed (Participants) | 39 | 39 | 40
  Serotype 23F | 33.3 [19.09 to 50.22] | 43.6 [27.81 to 60.38] | 32.5 [18.57 to 49.13]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 39 | 39 | 40
  Serotype 33F (non-Prevnar serotype) | 92.3 [79.13 to 98.38] | 87.2 [72.57 to 95.70] | 0.0 [0.00 to 8.81]

11. Secondary Outcome: Infants: Percentage of Participants With GMC ≥0.35 µg/mL at 1 Month After Vaccination 4
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: 1 month after Vaccination 4 (Month 11-15)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 52
Percentage of participants
  Serotype 1: number analyzed (Participants) | 32 | 35 | 36
  Serotype 1 | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 3: number analyzed (Participants) | 32 | 35 | 36
  Serotype 3 | 96.9 [83.78 to 99.92] | 97.1 [85.08 to 99.93] | 83.3 [67.19 to 93.63]
  Serotype 4: number analyzed (Participants) | 32 | 35 | 36
  Serotype 4 | 90.6 [74.98 to 98.02] | 97.1 [85.08 to 99.93] | 97.2 [85.47 to 99.93]
  Serotype 5: number analyzed (Participants) | 32 | 35 | 36
  Serotype 5 | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 6A: number analyzed (Participants) | 32 | 35 | 36
  Serotype 6A | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 6B: number analyzed (Participants) | 32 | 35 | 36
  Serotype 6B | 100.0 [89.11 to 100.0] | 97.1 [85.08 to 99.93] | 100.0 [90.26 to 100.00]
  Serotype 7F: number analyzed (Participants) | 32 | 35 | 36
  Serotype 7F | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 9V: number analyzed (Participants) | 32 | 35 | 36
  Serotype 9V | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 14: number analyzed (Participants) | 32 | 35 | 36
  Serotype 14 | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 97.2 [85.47 to 99.93]
  Serotype 18C: number analyzed (Participants) | 32 | 35 | 36
  Serotype 18C | 100.0 [89.11 to 100.00] | 97.1 [85.08 to 99.93] | 100.0 [90.26 to 100.00]
  Serotype 19A: number analyzed (Participants) | 32 | 35 | 36
  Serotype 19A | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 19F: number analyzed (Participants) | 32 | 35 | 36
  Serotype 19F | 100.0 [89.11 to 100.00] | 97.1 [85.08 to 99.93] | 100.0 [90.26 to 100.00]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 32 | 35 | 36
  Serotype 22F (non-Prevnar serotype) | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 5.6 [0.68 to 18.66]
  Serotype 23F | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 100.0 [90.26 to 100.00]
  Serotype 33F (non-Prevnar serotype) | 100.0 [89.11 to 100.00] | 100.0 [90.00 to 100.00] | 0.0 [0.00 to 9.74]

12. Secondary Outcome: Infants: Geometric Mean Concentration of Pneumococcal Serotype IgG Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: Before Vaccination 4 (Month 10-13)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 52
µg/mL
  Serotype 1: number analyzed (Participants) | 39 | 39 | 40
  Serotype 1 | 0.27 [0.22 to 0.33] | 0.30 [0.24 to 0.37] | 0.40 [0.31 to 0.51]
  Serotype 3: number analyzed (Participants) | 39 | 39 | 40
  Serotype 3 | 0.14 [0.11 to 0.18] | 0.21 [0.17 to 0.26] | 0.09 [0.07 to 0.12]
  Serotype 4: number analyzed (Participants) | 39 | 39 | 40
  Serotype 4 | 0.21 [0.17 to 0.25] | 0.26 [0.22 to 0.30] | 0.23 [0.18 to 0.30]
  Serotype 5: number analyzed (Participants) | 39 | 39 | 40
  Serotype 5 | 0.42 [0.35 to 0.49] | 0.40 [0.33 to 0.49] | 0.59 [0.44 to 0.79]
  Serotype 6A: number analyzed (Participants) | 39 | 39 | 40
  Serotype 6A | 0.35 [0.26 to 0.45] | 0.33 [0.26 to 0.42] | 0.63 [0.46 to 0.87]
  Serotype 6B: number analyzed (Participants) | 39 | 39 | 40
  Serotype 6B | 0.52 [0.41 to 0.66] | 0.50 [0.38 to 0.65] | 0.43 [0.30 to 0.62]
  Serotype 7F: number analyzed (Participants) | 39 | 39 | 40
  Serotype 7F | 0.56 [0.46 to 0.67] | 0.79 [0.66 to 0.94] | 0.89 [0.68 to 1.18]
  Serotype 9V: number analyzed (Participants) | 39 | 39 | 40
  Serotype 9V | 0.34 [0.29 to 0.40] | 0.42 [0.33 to 0.53] | 0.35 [0.27 to 0.47]
  Serotype 14: number analyzed (Participants) | 39 | 39 | 40
  Serotype 14 | 0.83 [0.62 to 1.11] | 0.92 [0.72 to 1.18] | 1.53 [1.13 to 2.07]
  Serotype 18C: number analyzed (Participants) | 39 | 39 | 40
  Serotype 18C | 0.16 [0.13 to 0.19] | 0.20 [0.16 to 0.25] | 0.28 [0.21 to 0.37]
  Serotype 19A: number analyzed (Participants) | 39 | 39 | 40
  Serotype 19A | 0.27 [0.21 to 0.35] | 0.32 [0.24 to 0.44] | 0.39 [0.31 to 0.50]
  Serotype 19F: number analyzed (Participants) | 39 | 39 | 40
  Serotype 19F | 0.28 [0.23 to 0.35] | 0.35 [0.29 to 0.43] | 0.48 [0.36 to 0.63]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 39 | 39 | 40
  Serotype 22F (non-Prevnar serotype) | 0.97 [0.82 to 1.16] | 1.14 [0.93 to 1.40] | 0.06 [0.05 to 0.07]
  Serotype 23F: number analyzed (Participants) | 39 | 39 | 40
  Serotype 23F | 0.23 [0.18 to 0.30] | 0.26 [0.19 to 0.35] | 0.26 [0.19 to 0.35]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 39 | 39 | 40
  Serotype 33F (non-Prevnar serotype) | 0.91 [0.75 to 1.10] | 0.96 [0.70 to 1.33] | 0.05 [0.05 to 0.05]

13. Secondary Outcome: Infants: Geometric Mean Concentration of Pneumococcal Serotype IgG Antibodies
Description: Pneumococcal serotype-specific IgG was measured in serum using an electrochemiluminescence assay.
Time Frame: 1 month after Vaccination 4 (Month 11-15)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infants: V114 Medium Dose | Infants: V114 High Dose | Infants: Prevnar 13™
Number analyzed (Participants) | 50 | 50 | 52
µg/mL
  Serotype 1: number analyzed (Participants) | 32 | 35 | 36
  Serotype 1 | 1.74 [1.33 to 2.29] | 2.32 [1.76 to 3.05] | 2.05 [1.58 to 2.66]
  Serotype 3: number analyzed (Participants) | 32 | 35 | 36
  Serotype 3 | 1.02 [0.84 to 1.24] | 1.26 [0.96 to 1.65] | 0.87 [0.65 to 1.17]
  Serotype 4: number analyzed (Participants) | 32 | 35 | 36
  Serotype 4 | 1.35 [0.99 to 1.84] | 1.84 [1.33 to 2.56] | 1.68 [1.25 to 2.25]
  Serotype 5: number analyzed (Participants) | 32 | 35 | 36
  Serotype 5 | 2.33 [1.80 to 3.00] | 2.53 [1.95 to 3.27] | 3.80 [2.80 to 5.17]
  Serotype 6A: number analyzed (Participants) | 32 | 35 | 36
  Serotype 6A | 5.59 [4.15 to 7.52] | 5.24 [3.81 to 7.19] | 9.13 [7.31 to 11.41]
  Serotype 6B: number analyzed (Participants) | 32 | 35 | 36
  Serotype 6B | 6.46 [5.20 to 8.01] | 5.12 [3.55 to 7.39] | 6.80 [5.38 to 8.60]
  Serotype 7F: number analyzed (Participants) | 32 | 35 | 36
  Serotype 7F | 2.94 [2.28 to 3.79] | 4.34 [3.49 to 5.40] | 5.26 [4.01 to 6.90]
  Serotype 9V: number analyzed (Participants) | 32 | 35 | 36
  Serotype 9V | 2.53 [1.85 to 3.47] | 2.36 [1.91 to 2.92] | 3.09 [2.39 to 4.00]
  Serotype 14: number analyzed (Participants) | 32 | 35 | 36
  Serotype 14 | 5.87 [4.05 to 8.52] | 4.42 [3.41 to 5.73] | 5.68 [4.08 to 7.92]
  Serotype 18C: number analyzed (Participants) | 32 | 35 | 36
  Serotype 18C | 1.68 [1.30 to 2.16] | 2.49 [1.90 to 3.27] | 2.62 [2.06 to 3.34]
  Serotype 19A: number analyzed (Participants) | 32 | 35 | 36
  Serotype 19A | 4.85 [3.62 to 6.50] | 4.92 [3.66 to 6.61] | 6.60 [5.23 to 8.34]
  Serotype 19F: number analyzed (Participants) | 32 | 35 | 36
  Serotype 19F | 4.24 [3.22 to 5.58] | 4.30 [3.15 to 5.87] | 4.28 [3.34 to 5.49]
  Serotype 22F (non-Prevnar serotype): number analyzed (Participants) | 32 | 35 | 36
  Serotype 22F (non-Prevnar serotype) | 6.57 [5.09 to 8.47] | 8.20 [6.61 to 10.17] | 0.07 [0.05 to 0.09]
  Serotype 23F: number analyzed (Participants) | 32 | 35 | 36
  Serotype 23F | 2.76 [2.11 to 3.61] | 2.99 [2.18 to 4.10] | 3.81 [2.89 to 5.01]
  Serotype 33F (non-Prevnar serotype): number analyzed (Participants) | 32 | 35 | 36
  Serotype 33F (non-Prevnar serotype) | 5.22 [3.87 to 7.04] | 4.84 [3.81 to 6.15] | 0.05 [0.05 to 0.06]

ADVERSE EVENTS:
Time Frame: Adults: all AEs: up to 14 days after vaccination; SAEs: up to 6 weeks after vaccination; infants: All AEs: up to 14 days after any vaccination; SAEs: up to 6 weeks after Vaccination 4.
Description: The analysis population included all randomized participants who received at least one dose of study vaccination. One cross-treated participant in the Infants: V114 Medium Dose + ACP group was excluded from the safety analysis.
Groups:
- V114 Medium Adults: Adult participants received a single 0.5 mL intramuscular injection of medium-dose V114 on Day 1
- V114 High Adults: Adult participants received a single 0.5 mL intramuscular injection of high-dose V114 on Day 1
- V114 Medium + ACP Adults: Adult participants received a single 0.5 mL intramuscular injection of medium-dose V114 with alternative carrier protein (ACP) on Day 1
- V114 High + ACP Adults: Adult participants received a single 0.5 mL intramuscular injection of high-dose V114 with ACP on Day 1
- V114 Medium Infants: Infant participants received a single 0.5 mL intramuscular injection of medium-dose V114 at 2, 4, 6, and 12-15 months of age
- V114 High Infants: Infant participants received a single 0.5 mL intramuscular injection of high-dose V114 at 2, 4, 6, and 12-15 months of age
- V114 Medium + ACP Infants: Infant participants received a single 0.5 mL intramuscular injection of medium-dose V114 with ACP at 2, 4, 6, and 12-15 months of age
- V114 High + ACP Infants: Infant participants received a single 0.5 mL intramuscular injection of high-dose V114 with ACP at 2, 4, 6, and 12-15 months of age
- Prevnar 13 Infants: Infant participants received a single 0.5 mL intramuscular injection of Prevnar 13™ at 2, 4, 6, and 12-15 months of age
Arm/Group | V114 Medium Adults | V114 High Adults | V114 Medium + ACP Adults | V114 High + ACP Adults | V114 Medium Infants | V114 High Infants | V114 Medium + ACP Infants | V114 High + ACP Infants | Prevnar 13 Infants
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/50 | 0/50 | 0/51 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 5/50 | 4/50 | 1/51 | 3/52 | 4/52
Other Adverse Events (participants affected / at risk) | 18/20 | 19/20 | 19/20 | 18/20 | 47/50 | 46/50 | 49/51 | 51/52 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Medium Adults (N=20) | V114 High Adults (N=20) | V114 Medium + ACP Adults (N=20) | V114 High + ACP Adults (N=20) | V114 Medium Infants (N=50) | V114 High Infants (N=50) | V114 Medium + ACP Infants (N=51) | V114 High + ACP Infants (N=52) | Prevnar 13 Infants (N=52)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Child maltreatment syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal insufficient breast milk syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Medium Adults (N=20) | V114 High Adults (N=20) | V114 Medium + ACP Adults (N=20) | V114 High + ACP Adults (N=20) | V114 Medium Infants (N=50) | V114 High Infants (N=50) | V114 Medium + ACP Infants (N=51) | V114 High + ACP Infants (N=52) | Prevnar 13 Infants (N=52)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 3 (4) | 4 (4) | 1 (2) | 6 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (4) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (8) | 4 (4) | 2 (2) | 5 (5)
Fatigue (General disorders) | 7 (8) | 9 (9) | 9 (9) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 5 (5) | 2 (2) | 2 (2) | 19 (27) | 21 (34) | 16 (27) | 17 (31) | 15 (26)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 19 (26) | 18 (31) | 15 (18) | 19 (38) | 13 (28)
Injection site pain (General disorders) | 17 (20) | 19 (23) | 18 (24) | 17 (21) | 32 (69) | 31 (67) | 22 (39) | 38 (82) | 21 (46)
Injection site swelling (General disorders) | 5 (5) | 6 (6) | 4 (4) | 5 (5) | 10 (13) | 16 (23) | 10 (18) | 19 (30) | 13 (19)
Injection site warmth (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 17 (28) | 14 (26) | 16 (23) | 16 (25) | 21 (37)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 5 (6)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 0 (0) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 4 (4) | 7 (8) | 3 (3) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 16 (34) | 24 (40) | 16 (28) | 27 (55) | 24 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10) | 7 (7) | 10 (11) | 2 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 30 (69) | 34 (76) | 31 (91) | 38 (97) | 39 (95)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 41 (143) | 41 (167) | 46 (195) | 47 (200) | 44 (171)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 5 (6) | 1 (1) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 3 (4) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 1 (1) | 4 (4)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT02531373/Prot_SAP_000.pdf